CLINICAL TRIAL: NCT03308409
Title: Clinical Randomized Multicentric Trial to Evaluate the Comparative Effectiveness and Safety of Three Protocols Using Low-intensity Shock Waves for the Treatment of Erectile Dysfunction
Brief Title: Comparative Effectiveness and Safety of Three Protocols Usin Li-ESWT for Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMGC-3
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Patients who met the selection criteria were randomly assigned to one of three groups: weekly protocol, monthly protocol, or booster protocol, in a 1:1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Protocol 1 (Active Comparator): Low-intensity extracorporeal shock wave therapy (Li-ESWT): Six sessions, one per week, with 3000 pulses at 0.20 mj/mm2, at a frequency of 4Hz. At all of the shockwave sessions, 2000 pulses will be distributed to the body of the penis and 1000 pulses will be applied to the base.
  Interventions: Other: Low-intensity extracorporeal shock wave therapy (Li-ESWT)
- Protocol 2 (Experimental): Low-intensity extracorporeal shock wave therapy (Li-ESWT): Six initial sessions, one per week, with 3000 pulses at 0.20 mj/mm2, at a frequency of 4Hz for six weeks, followed by monthly maintenance sessions (every 4 weeks) for five months. At all of the shockwave sessions, 2000 pulses will be distributed to the body of the penis and 1000 pulses will be applied to the base.
  Interventions: Other: Low-intensity extracorporeal shock wave therapy (Li-ESWT)
- Protocol 3 (Experimental): Low-intensity extracorporeal shock wave therapy (Li-ESWT): Six monthly sessions in which 3000 pulses will be applied at 0.20 mj/mm2, at a frequency of 4Hz, with 2000 pulses distributed to the body of the penis and 1000 pulses applied to the base
  Interventions: Other: Low-intensity extracorporeal shock wave therapy (Li-ESWT)

INTERVENTIONS:
Other: Low-intensity extracorporeal shock wave therapy (Li-ESWT) — Low-intensity shock waves are acoustic wavelengths which are transmitted continuously at a frequency between 16 and 20 megahertz for under 10 microseconds. They generate a pressure pulse and transport energy as they propagate through a medium. Three different methods can be used to generate this type of wave: electro-hydraulics, electro-magnetics and piezoelectricity. Regardless of the method, when the shock waves are applied to an organ they interact with the deep tissue. This causes stress and small mechanical traumas, activating the release of angiogenic factors which induce new vascularization of the affected tissue, thereby improving blood flow.

SUMMARY:
The patients with primary erectile dysfunction (IIEF-EF <26 points), will be randomly assigned to three shockwave treatment protocols: Protocol 1 six sessions, one per week; Protocol 2, six initial sessions, one per week, followed by monthly maintenance sessions (every 4 weeks) for five months; Protocol 3, six monthly sessions. The EHS and IIEF-EF scores will be compared as well as the possible adverse events from the therapy upon beginning and completing the treatment and at the 3-month and 6-month follow-ups. Self-esteem and quality of life will also be evaluated using the SEAR scale.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years of age
* Presence of ED for more than 3 months in over 50% of sexual intercourses.
* Baseline ED domain score under 26 on the IIEF-15 EF domain.
* Patient agrees to participate in the trial by providing signed informed consent.

Exclusion Criteria:

* EHS score of 4.
* Patients with an INR over 3.
* Patients with sickle-cell anemia.
* Patients with clinical suspicion of hypogonadism (AMS over 36).
* Endocrine diseases that present with ED, such as acromegaly, gigantism, Addison's disease, hyperprolactinemia, androgen deficiency.
* Active vesicular, prostrate or colon cancer.
* Radical prostatectomy or other radical pelvic surgery.
* History of pelvic radiation therapy.
* Patients with ED of psychological origin.
* Spinal cord injury or other neurological diseases associated with ED.
* Anatomical penile dysfunction, penile implant.
* Patients with active infections or lesions on the penis or pubic area.
* Patients with ED secondary to drug therapy (antiandrogen therapy, alpha blockers for BPH, use of corticosteroids, medication for Parkinson's disease, antipsychotics).
* Abuse of psychoactive substances.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
IIEF-EF score 6 months after completing the treatment | 6 month follow-ups
  This is a highly sensitive and specific scale for detecting changes in erectile function in response to treatment. The degree of dysfunction is scored on a range of 0 to 30 points on the Erectile Functioning domain (questions 1, 2, 3, 4, 5, 15). The categories are: severe between 0 and 10, moderate between 11 and 16, mild-to-moderate between 17 and 21, mild between 22 and 25, and no ED between 26 and 30.

SECONDARY OUTCOMES:
Erection Hardness Score | 3-month and 6-month follow-ups
  The EHS has a single Likert scale: 0 = Penis does not increase in size; 1= the penis increases in size but is not hard; 2 = the penis is hard but not hard enough for penetration; 3 = the penis is hard enough for penetration but not completely hard; 4 = the penis is completely hard and fully rigid
Clinical improvement | 6-month follow-ups
  For patients with moderate ED, a 5-point increase in the IIEF-EF score is considered improvement. For patients with mild ED a 2-point increase on this scale is considered improvement. And for those with severe ED a 7-point change is considered improvement.
Number of satisfactory relations | 3-month and 6-month follow-ups
  According to the patient's journal records. For the purpose of this study, satisfactory relations are defined as the increase in rigidity and duration of the erection as evaluated by the patient and his partner. For patients who were not able to penetrate before treatment, satisfactory relations will include not only an increase in rigidity and duration of the erection but also the ability to penetrate.

CONTACTS AND LOCATIONS:
Locations (2):
- Boston Medical Group Colombia, Bogotá, Cundinamarca, Colombia
- Boston Medical Group, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No